CLINICAL TRIAL: NCT01876199
Title: Targeted Screening of At-Risk Adults for Acute HIV-1 Infection
Acronym: AHI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: International AIDS Vaccine Initiative (Network); KEMRI-Wellcome Trust Collaborative Research Program (Other); University of Washington (Other); Kenya Ministry of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SSC2359; 167-12 (Other: OXTREC)
Record Dates: First submitted 2013-06-10; First posted 2013-06-12 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-08

CONDITIONS: HIV
Keywords: HIV-1; acute; diagnosis; pharmacies; healthcare facilities
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intense follow up (Experimental): 2-week follow up appointment with addition of a reminder mobile phone call or short text message (SMS) if possible, plus a home visit by a community counselor if the participant fails to present on the appointed date.
  Interventions: Behavioral: intense follow up
- standard follow-up (No Intervention): 2-week follow-up appointment with no reminders

INTERVENTIONS:
Behavioral: intense follow up
  Arms: Intense follow up

SUMMARY:
In this research, the investigators want to see if early detection of HIV infection can be improved by testing young adults who seek urgent health care from pharmacies and healthcare facilities with symptoms similar to those people get with recent HIV infection.

Specific objectives:

1. What proportion of people presenting with these symptoms are HIV positive at the point of seeking urgent health care?
2. What proportion of those who test negative or where the result is unclear (one rapid test positive and one negative) at first rapid HIV testing, will test positive two weeks later?
3. What is the best way (SMS, phone call or home visit) to remind people to come for the second test after two weeks?
4. Will young adults who seek urgent health care for fever, body pains, diarrhoea or an STD from pharmacies or health facilities find it acceptable to be invited for an HIV-1 test at the time of health care seeking?

Hypotheses

1. Targeted screening for AHI among patients seeking health care for symptoms compatible with AHI or sexually transmitted disease (STD) will identify AHI cases in more than 1% of those screened.
2. Intense follow-up of patients evaluated for AHI will improve rates of repeat HIV-1 testing 2-4 weeks after initial health-care seeking, relative to standard practice (i.e., recommendation to return for testing on a given date).

ELIGIBILITY:
Inclusion Criteria:

* symptom score of 2 or more: Confirmed fever (≥37.5 °C axillary), reported diarrhoea, or evidence of STD (variable score=2); reported body pains, or report of more than one sexual partners in past 2 months (variable score=1)
* resident in Mtwapa or Shanzu or planning to stay in Mtwapa for approximately 4 weeks duration
* willing to give locator information (including mobile phone number)
* negative or unknown HIV status

Exclusion Criteria:

* patients not meeting inclusion criteria

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 522 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Difference in Number and proportion of adults responding to standard appointment versus intense follow up. | 2 weeks

SECONDARY OUTCOMES:
Number and proportion of adults diagnosed with AHI by rapid antibody seroconversion. | 2 weeks

OTHER OUTCOMES:
Number and proportion of adults diagnosed with AHI by p24 antigen testing alone | 2 weeks
Proportion of patients diagnosed with AHI who successfully enroll in HIV-1 care | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- KEMRI Mtwapa, Kilifi, Kenya

REFERENCES:
- [Derived] Mugo PM, Wahome EW, Gichuru EN, Mwashigadi GM, Thiong'o AN, Prins HA, Rinke de Wit TF, Graham SM, Sanders EJ. Effect of Text Message, Phone Call, and In-Person Appointment Reminders on Uptake of Repeat HIV Testing among Outpatients Screened for Acute HIV Infection in Kenya: A Randomized Controlled Trial. PLoS One. 2016 Apr 14;11(4):e0153612. doi: 10.1371/journal.pone.0153612. eCollection 2016. PMID 27077745
- See also: KEMRI Wellcome Trust Research Programme — http://www.kemri-wellcome.org
- See also: KEMRI Wellcome on SiteFinder — https://sitefinder.tghn.org/sites/kemri-wellcome-trust-research-programme/